CLINICAL TRIAL: NCT03316339
Title: Effect of Opioid-free Anesthesia on Postoperative Opioid-related Adverse Events After Major or Intermediate Non-cardiac Surgery: a Multicenter Prospective Randomized Controlled Study
Brief Title: Postoperative and Opioid Free Anesthesia
Acronym: POFA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35RC16_9842_POFA
Record Dates: First submitted 2017-10-13; First posted 2017-10-20 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia; Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Control (Active Comparator)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Opioid-free anesthesia
  Arms: Dexmedetomidine
Drug: Remifentanil — Opioid anesthesia
  Arms: Control

SUMMARY:
Since the 1960's, intraoperative administration of opioids is considered a keystone of anesthesia as well as hypnotics and muscle relaxants. Synthetic opioids were introduced to achieve hemodynamic stability during anesthesia. They allow an inhibition of the sympathetic system without cardiovascular collapse and histamine release. Since then, anesthesia has changed from inhalation to multimodal anesthesia with lower doses of hypnotic. In 2017, the intraoperative objectives of hypnosis, hemodynamic stability, immobility and anticipation of postoperative analgesia can be achieved without opioids. Moreover, opioid administration consequences are neither scarce nor benign for the patient. Perioperative opioids are associated with nausea and vomiting, sedation, ileus, confusion/delirium, respiratory depression, increased postoperative pain and morphine consumption, immunodepression, hyperalgesia and chronic postoperative pain. Among these complications, hypoxemia, ileus and confusion/delirium are the most frequent.

Efficacious multimodal analgesia and anesthesia are the basis of successful fast-track surgery. These multidrug regimens aim at decreasing postoperative pain, intra- and postoperative opioid requirements, and subsequently, opioid-related adverse effects and to fasten recovery. Opioid-free postoperative analgesia has been recommended for more than 10 years. Opioid-free anesthesia (OFA) is based on the idea that hemodynamic stability can be achieved without opioids during anesthesia. OFA is multimodal anesthesia associating hypnotics, N-methyl-D-aspartate (NMDA) antagonists, local anesthetics, anti-inflammatory drugs and alpha-2 agonists (Dexmedetomidine).

Proofs of the effect of OFA on reducing opioid-related adverse effects after major or intermediate non-cardiac surgery are still scarce. We hypothesized that the reduced opioid consumption during and after surgery allowed by OFA compared with standard of care will be associated with a reduction of postoperative opioid-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a scheduled major or intermediate non-cardiac surgery,
* Benefiting from the health insurance system,
* Having signed an informed consent.

Exclusion Criteria:

* Pregnant or breast feeding women,
* Allergy to dexmedetomidine or one of its excipients,
* Allergy to one of the drugs used for anesthesia or one of their excipients,
* Urgent surgery,
* Intracranial surgery,
* Transplant surgery or transplanted patients,
* Surgery with planned regional anesthesia,
* Outpatient surgery,
* Atrioventricular block, intraventricular or sinoatrial block,
* Treatment by chronic betablockers and HR < 50 bpm,
* Heart failure with LVEF < 40%,
* Adam-Stokes syndrome,
* Epilepsy or seizures,
* Uncontrolled hypotension,
* Acute cerebral pathology,
* Obstructive sleep apnea syndrome,
* Severe hepatic insufficiency (Prothrombin Ratio < 15%),
* Patients in whom the CAM-ICU cannot be performed (deaf patients for example)
* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Occurence of a severe postoperative opioid-related adverse event defined as : postoperative hypoxemia or postoperative ileus (POI) or postoperative cognitive dysfunction (POCD). | Within the first 48 hours after extubation
  Postoperative hypoxemia is defined as an oxygen saturation (SpO2) < 95% with a need for oxygen supplementation within the first 48h after extubation; the duration of oxygen treatment will also be recorded.
  Postoperative ileus is defined as an absence of flatus or stools within the first 48h after extubation.
  Postoperative cognitive dysfunction will be evaluated using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) by a care provider (either anesthesiologist or nurse).

SECONDARY OUTCOMES:
Number of episodes of postoperative pain (numeric rating scale ≥ 3), at rest | Within 48 hours after extubation
Opioid consumption | During the 48 hours following extubation
Time between the end of remifentanil or dexmedetomidine administration and an Aldrete score > 9 (when applicable) | Within 48 hours after extubation
Time between the end of remifentanil or dexmedetomidine administration and extubation | Hour 0 = extubation
Rate of unscheduled admission in intensive care unit | Within 48 hours after extubation
Number of postoperative nausea and vomiting (PONV) episodes | During the 48 hours following extubation
Hospital length of stay (max 28 days) defined as the number of days after extubation before first hospital discharge | Day 28
Number of bradycardia, hypotension and hypertension events during surgery and number of rescue medications during surgery | During surgery (maximum duration of 7 hours)
  Bradycardia is defined as the number of episodes with atropine administration. Hypotension is defined as mean arterial blood pressure < 65 mmHg. Hypertension is defined as mean arterial blood pressure > 90 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BELOEIL, Principal Investigator — Rennes University Hospital
Locations (11):
- France (11):
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Beaujon Hospital, Clichy
  - Lille University Hospital, Lille
  - Metz-Thionville Hospital, Metz
  - Montpellier University Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - Nimes University Hospital, Nîmes
  - Perigueux Hospital, Périgueux
  - Rennes University Hospital, Rennes
  - Saint-Brieuc Hospital, Saint-Brieuc
  - Toulouse University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beloeil H, Laviolle B, Menard C, Paugam-Burtz C, Garot M, Asehnoune K, Minville V, Cuvillon P, Oger S, Nadaud J, Lecoeur S, Chanques G, Futier E; SFAR research network. POFA trial study protocol: a multicentre, double-blind, randomised, controlled clinical trial comparing opioid-free versus opioid anaesthesia on postoperative opioid-related adverse events after major or intermediate non-cardiac surgery. BMJ Open. 2018 Jun 30;8(6):e020873. doi: 10.1136/bmjopen-2017-020873. PMID 29961015